CLINICAL TRIAL: NCT03435601
Title: A Randomised, Double-blind, Placebo-controlled Phase II Study to Target the Type I IFN Receptor by Administrating Anifrolumab in RA Patients With a High IFN Signature (TarIFNiRA)
Brief Title: A Study to Target the Type I IFN Receptor by Administrating Anifrolumab in RA Patients With a High IFN Signature (TarIFNiRA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josef Smolen, Univ. Prof. Dr. (Other)
Responsible Party: Sponsor-Investigator, Josef Smolen, Univ. Prof. Dr., Sponsor-Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TarIFNiRA; 2017-001717-92 (EudraCT Number)
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; IFN-Signature; Anifrolumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (Experimental): Anifrolumab 300 mg IV administration Q4W, a total of 6 doses
  Interventions: Drug: Anifrolumab
- Placebo (Placebo Comparator): Placebo IV administration Q4W, a total of 6 doses
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Anifrolumab — IV Administration of Anifrolumab 300 mg every 4 weeks from week 0 to week 20 for a total of 6 doses.
  At week 24 patients will continue the current study for another 8 weeks to complete a 12-week safety follow-up after the last dose of investigational products (last dose of investigational product will be given at week 20).
  The total study duration could be up to approximately 36 weeks (including the screening period).
  Arms: Anifrolumab
Drug: Placebos — Placebo IV administration Q4W, a total of 6 doses At week 24 patients will continue the current study for another 8 weeks to complete a 12-week safety follow-up after the last dose of investigational products (last dose of investigational product will be given at week 20).
  The total study duration could be up to approximately 36 weeks (including the screening period).
  Arms: Placebo

SUMMARY:
A multicenter, randomised, double-blind, placebo-controlled Phase 2A/ proof-of-concept study to evaluate the efficacy and safety of an intravenous treatment regimen of 300 mg Anifrolumab versus placebo in patients with moderately to severely active RA who did not respond to biological disease-modifying anti-rheumatic drugs (bDMARDs) and who have a high type I IFN gene signature.

DETAILED DESCRIPTION:
Background: Rheumatoid arthritis (RA) is the most common chronic inflammatory joint disorder with a prevalence of about 0.5-1% and results in joint inflammation and damage, which causes loss-of-function and disability, and ultimately results in loss of labour participation, loss of independence in daily life and high societal costs. Conventional synthetic DMARDs (csDMARDs), especially methotrexate, represent the first-line treatment in RA. If, however, the treatment target is not achieved with the first DMARD strategy escalation in the treatment regimen is needed. The current praxis is to add a biological (b) DMARD (e.g. TNF inhibitors, TNFi). With the growing evidence that type I IFNs play an important role in RA, inhibition of the biological activity of type I IFNs with anifrolumab may be a novel efficacious therapy for the treatment of RA and its significant unmet medical need.

Objective: To evaluate the efficacy of Anifrolumab compared to placebo on RA disease activity in patients with an increased type I IFN gene signature

Methods: This is a Phase 2A (proof-of-concept), multicenter, randomised, double-blind, placebo-controlled pilot study, to evaluate the efficacy and safety of an intravenous treatment regimen of 300 mg Anifrolumab versus placebo. Patients with moderately to severely active RA who did not respond to at least one TNFi but who had not more than three bDMARDs and who also have a high IFN- transcript score will be included.

Expected Results: The hypothesis underlying this protocol is that blocking type I IFN signaling through the human type I IFN receptor with Anifrolumab will reduce the severity of disease in RA patients, who have an activated type I IFN response.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 through 70 years at the time of screening
* Written informed consent
* Weigh ≥50.0 kg and ≤100.0 kg at screening
* Diagnosis of RA according to the 2010 ACR/EULAR classification criteria for RA
* At study entry, patients must take at least one conventional synthetic (cs)DMARD (methotrexate (MTX), leflunomide, sulfasalazine (SSZ)) regularly for at least the preceding 12 weeks, with stable doses for at least the preceding 8 weeks.
* moderately to severely active RA: ≥4 tender joints of 28 joints examined, ≥4 swollen joints of 28 joints examined and an elevated serum C-reactive protein level (CRP).
* Received at least one TNF-inhibitor (TNFi) but not more than 3 biological (b)DMARDs and discontinued treatment because of an insufficient response after at least 3 months.
* Oral Glucocorticoids (OCS) are allowed at stable doses of ≤10 mg/day prednisone or equivalent, if already used before the screening visit, dose must be stable for at least 2 weeks, and will be kept stable throughout the course of the study
* High type I IFN gene signature test
* Seronegative for human immunodeficiency virus (HIV) and negative test for hepatitis B surface antigen and hepatitis C - antibodies
* Negative serum β-human chorionic gonadotropin (β-hCG) test at screening (females of childbearing potential only).
* Females of childbearing potential must use 2 effective methods of avoiding pregnancy, only one of which is a barrier method, from screening until 12 weeks after the final dose of the investigational product unless the subject is surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy), has a sterile male partner, is 1 year post-menopausal, or practices sustained abstinence.Cessation of birth control after the specified period for investigational product should be discussed with a responsible physician. Post-menopausal is defined as at least 1 year since last menses and the subject having an elevated follicle- stimulating hormone (FSH) level greater than the central laboratory value of post-menopausal at screening
* All males (sterilised or non-sterilised) who are sexually active must use condom (with spermicide where commercially available for contraception if sexually active with a woman of child bearing potential) from Day 0 until at least 12 weeks after receipt of the final dose of the investigational product. It is strongly recommended that female partners of child bearing potential of male subjects also use a highly effective method of contraception (other than a barrier method) throughout this period.
* Male subjects must not donate sperm during the course of the study and for 12 weeks after the last dose of the investigational product.
* Females with an intact cervix must have documentation of a normal Pap smear with no documented malignancy (e.g., cervical intraepithelial neoplasia grade III [CIN III], carcinoma in situ [CIS], or adenocarcinoma in situ [AIS]) within 2 years prior to randomization. Any abnormal Pap smear result documented within 2 years prior to randomization must be repeated to confirm patient eligibility.
* Meets all of the following tuberculosis (TB) criteria:

  * No history of latent or active TB prior to screening, with the exception of latent TB with documented completion of appropriate treatment
  * No signs or symptoms suggestive of active TB from medical history or physical examination
  * No recent contact with a person with active TB OR if there has been such contact, referral to a physician specialising in TB to undergo additional evaluation prior to randomisation (documented appropriately in source), and, if warranted, receipt of appropriate treatment for latent TB at or before the first administration of investigational product
  * Negative QuantiFERON-tuberculosis Gold [QFT-G] test for tuberculosis within 3 months prior to randomisation
* A chest radiograph with no evidence of current active infection (eg, tuberculosis) or old active TB, malignancy, or clinically significant abnormalities obtained during the screening period or anytime within 12 weeks prior to signing of the informed consent

General Exclusion criteria:

* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of patient safety or study results
* Concurrent enrolment in another clinical study with an investigational product
* Individuals involved with the conduct of the study, their employees, or immediate family members of such individuals
* Lactating or pregnant females or females who intend to become pregnant anytime from initiation of screening until the 12-week safety follow-up period following last dose of investigational product
* Current alcohol, drug or chemical abuse, or a history of such abuse within 1 year before Week 0 (Day 0)
* Major surgery within 8 weeks before signing informed consent form (ICF) or elective major surgery planned during the study period
* Spontaneous or induced abortion, still or live birth, or pregnancy ≤4 weeks prior to signing the ICF
* Low type I IFN transcript scores in peripheral whole blood (type I Interferon Gene signature test)
* At screening (within 4 weeks before Week 0 [Day 0]), any of the following:
* Aspartate aminotransferase (AST) >2.0 × upper limit of normal (ULN)
* Alanine aminotransferase (ALT) >2.0 × ULN
* Total bilirubin >ULN (unless due to Gilbert's syndrome)
* Serum creatinine >2.0 mg/dL (or >181 μmol/L)
* Urine protein/creatinine ratio >2.0 mg/mg (or >226.30 mg/mmol)
* Neutrophil count <1000/μL (or <1.0 × 109/L)
* Platelet count <150.000/μL (or <150 × 109/L)
* Haemoglobin <8 g/dL (or <80 g/L)
* Glycosylated haemoglobin (HbA1c) >8% (or >0.08) at screening (diabetic patients only)

Exclusion criteria related to concomitant medications:

* Receipt of any investigational product (small molecule or biologic agent) within 4 weeks or 5 half-lives prior to signing of the ICF.
* Prior receipt of Anifrolumab
* Prior receipt of a JAK-inhibitor
* A known history of allergy or reaction to any component of the investigational product formulation or history of anaphylaxis to any human gamma globulin therapy
* Regular use of >1 nonsteroidal anti-inflammatory drug (NSAID) within 2 weeks prior to week 0 (Day 0); OR receipt of fluctuating doses of a NSAID within 2 weeks prior to Week 0 (Day 0)
* Receipt of any of the following: Intra-articular, intramuscular or intravenous glucocorticosteroids within 6 weeks prior to Day 0
* Any live or attenuated vaccine within 8 weeks prior to signing the ICF (administration of killed vaccines is acceptable); Patients should be up to date on required vaccinations, including influenza [inactivated/recombinant] vaccine prior to study entry
* Bacillus Calmette-Guerin (BCG) vaccine within 1 year of signing the informed consent form
* Blood transfusion within 4 weeks prior to signing the ICF

Exclusion criteria related to other diseases:

* History of any non-RA disease that has required treatment with oral or parenteral corticosteroids for more than a total of 2 weeks within the last 24 weeks prior to signing the ICF

Exclusion criteria related to infection and malignancy risk factors:

* Splenectomy
* Any severe herpes infection at any time prior to Week 0 (Day 0), including, but not limited to, disseminated herpes (ever), herpes encephalitis (ever), recurrent herpes zoster (defined as 2 episodes within 2 years) or ophthalmic herpes (ever)
* Any herpes zoster infection that has not completely resolved within 12 weeks prior to signing the ICF
* Opportunistic infection requiring hospitalisation or parenteral antimicrobial treatment within 3 years of randomisation
* Any of the following:

  * Clinically significant chronic infection (ie, osteomyelitis, bronchiectasis, etc) within 8 weeks prior to signing the ICF (chronic nail infections are allowed)
  * Any infection requiring hospitalisation or treatment with intravenous anti-infectives not completed at least 4 weeks prior to signing the ICF
* Any infection requiring oral anti-infectives (including antivirals) within 2 weeks prior to Day 0
* History of cancer, apart from:

  * Squamous or basal cell carcinoma of the skin treated with documented success of curative therapy ≥3 months prior to Week 0 (Day 0)
  * Cervical cancer in situ treated with apparent success with curative therapy ≥1 year prior to Week 0 (Day 0)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Achieving an ACR 20 response at week 24 | Week 24
  To evaluate the efficacy of Anifrolumab compared to placebo on RA disease activity in patients with an increased type I IFN gene signature

SECONDARY OUTCOMES:
Absolute and relative change in the Simplified Disease Activity Index (SDAI) after 24 weeks | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Absolute and relative change in Clinical Disease Activity Index (CDAI) at week 24 and at every visit before and after week 24 | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Absolute and relative change in Disease Activity Score 28 (DAS28) after 24 weeks | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Achieving a EULAR response (good, moderate) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Achieving a SDAI response (50%, 70%, 85%) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Achieving a CDAI response (50%, 70%, 85%) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Achieving an ACR response (20%, 50%, 70%) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Change in quality of life (SF-36) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Change in physical function (HAQ) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Change in pain (visual analog scale, VAS) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Change in fatigue (visual analog scale, VAS) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Change in sleep (visual analog scale, VAS) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Proportion achieving a low disease activity state (CDAI≤10, SDAI≤11) after 24 weeks | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Proportion achieving a remission state (CDAI≤2.8; SDAI≤3.3; ACR/EULAR Boolean) after 24 weeks | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Proportion achieving DAS28≤3.2 after 24 weeks | Week 24
  To evaluate the effect of Anifrolumab compared to placebo
Change in Kessler Psychological Distress Scale (K10) | Week 24
  To evaluate the effect of Anifrolumab compared to placebo K10 is used as a simple measure of psychological distress, involves 10 questions about emotional states with a 5-level response scale and ranges from "all of the time" to "none of the time"

OTHER OUTCOMES:
To evaluate the safety and tolerability of Anifrolumab, relative to placebo | Week 24
  To evaluate the safety and tolerability of Anifrolumab, relative to placebo in terms of occurence of adverse events (AE), including adverse events of special interest (AESI)
To evaluate the safety and tolerability of Anifrolumab, relative to placebo | Week 24
  To evaluate the safety and tolerability of Anifrolumab, relative to placebo in terms of changes from baseline in vital signs (e.g. blood pressure)
To evaluate the safety and tolerability of Anifrolumab, relative to placebo | Week 24
  To evaluate the safety and tolerability of Anifrolumab, relative to placebo in terms of safety laboratory results (blood chemistry, liver biochemistry,...)
Pharmacodynamics (PD) of Anifrolumab | Week 24, Week 28
  Anifrolumab serum / plasma levels (Elisa)
Anti-drug antibody levels (ADA, anti-Anifrolumab antibody levels) | Week 24, Week 28
  Anti-drug antibody levels will be measured by Elisa
To evaluate the effects of Anifrolumab on the peripheral blood transcriptome | Week 24
  To explore whether changes of the transcriptome can be used to monitor and/or predict treatment response
To evaluate the effects of Anifrolumab on the peripheral blood methylome | Week 24
  To explore whether the changes of the methylome can be used to monitor and/or predict treatment response

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medizinische Universität Graz, Klinische Abteilung für Rheumatologie und Immunologie, Graz
  - Medizinische Universität Wien, Innere Medizin III, Abteilung für Rheumatologie, Vienna
  - Krankenhaus Hietzing, 2. Medizinische Abteilung, Vienna